CLINICAL TRIAL: NCT04177147
Title: Primary Care Clinicians' Responses to a Hypoglycemia Risk Calculator for Diabetes Mellitus in Ambulatory Care
Acronym: HG_Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael Weiner, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Merck RI 22
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hypoglycemia; Diabetes Mellitus
Keywords: Hypoglycemia; Diabetes mellitus; Clinical decision support; Electronic health records
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Clinicians were randomized to see, or not see, a clinical decision-support alert tool when evaluating outpatients with diabetes mellitus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical decision support via alert tool (Experimental): Clinicians received access to the electronic alert tool, which automatically displayed patients' risk of hypoglycemia.
  Interventions: Other: Clinical decision support via alert tool
- Usual care (No Intervention): Clinicians did not receive access to the electronic alert tool.

INTERVENTIONS:
Other: Clinical decision support via alert tool — The alert tool displays the risk of hypoglycemia for outpatients with diabetes mellitus.
  Arms: Clinical decision support via alert tool

SUMMARY:
Hypoglycemia (HG) is common and can be dangerous in diabetes mellitus, so identifying patients at risk may lead to useful preventive strategies and improved quality of care and health outcomes. This study will test the implementation of a computerized alert tool for clinicians.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common non-communicable diseases worldwide and is a major cause of morbidity and mortality. An estimated 346 million people had diabetes in 2011, and diabetes is predicted to become the seventh leading cause of death in the world by the year 2030. In the United States, the incidence of diabetes nearly tripled between 1990 and 2010, with 1.9 million new cases diagnosed in 2010. Hypoglycemia (HG) is recognized as a limiting factor in optimal glycemic management of patients with diabetes. This potentially costly condition, occurring in approximately 20% to 60% of patients who receive oral medications for diabetes, threatens patient safety, quality of life, and potentially, cardiovascular health. Investigators have identified risk factors for HG, built a risk calculator for use by clinicians, integrated the calculator into the G3 electronic medical record system, and demonstrated our ability to collect data about outcomes. In this project, investigators studied the outcomes of implementing the risk calculator tool into clinical practice in ambulatory primary care. The findings and tools developed from this project will promote improved patient safety and medical care for diabetes.

ELIGIBILITY:
The study included clinicians who were scheduled to provide primary care during the four-month intervention period.

Inclusion Criteria for patients:

* Being at least 21 years of age
* Have been prescribed or dispensed a drug for diabetes mellitus

Exclusion Criteria for patients:

N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypoglycemia during the study period | Five-month follow-up period
  Participants with hypoglycemia had blood glucose level less than 70 mg/dL

SECONDARY OUTCOMES:
Number of participants with changes to prescriptions for diabetes or antibiotics: new, refilled, changed, or discontinued | Five-month follow-up period
  Prescriptions for insulin and sulfonylurea drugs are assessed

OTHER OUTCOMES:
Number of participants with inpatient or outpatient medical encounters | Five-month follow-up period
  Includes emergency encounters
Number of participants undergoing patient education related to diabetes | Five-month follow-up period
  Text analysis of medical encounter notes
Number of A1c, glucose, and creatinine blood tests | Five-month follow-up period
  Mean and SD

REFERENCES:
- [Derived] Weiner M, Cummins J, Raji A, Ofner S, Iglay K, Teal E, Li X, Engel SS, Knapp K, Rajpathak S, Baker J, Chatterjee AK, Radican L. A randomized study on the usefulness of an electronic outpatient hypoglycemia risk calculator for clinicians of patients with diabetes in a safety-net institution. Curr Med Res Opin. 2020 Apr;36(4):583-593. doi: 10.1080/03007995.2020.1717451. Epub 2020 Feb 6. PMID 31951747